CLINICAL TRIAL: NCT06883019
Title: A Real World Study of Lecanemab Treatment in Participants with Early Onset Familial Alzheimer's Disease
Brief Title: Lecanemab for Early Onset Familial Alzheimer's Disease
Status: Recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Wang Gang, Professor, RenJi Hospital
Other Study IDs: LEOFAD-01
Record Dates: First submitted 2025-03-12; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to learn about the efficacy of Lecanemab treatment for early-onset familial Alzheimer's disease (AD) in patients under 65 years of age with a family history of AD. Participants will receive Lecanemab at a dosage of 10 mg/kg every two weeks for a total of 18 months and will undergo cognitive assessments, PET and MRI scans, blood/fluid tests and whole genome sequencing. The study will explore the effects of genetic and hereditary factors on the efficacy of Lecanemab treatment in early-onset familial AD patients.

ELIGIBILITY:
Inclusion Criteria:

* Age at onset ≤ 65 years, with a minimum age of 18 years; no restriction on gender.
* Diagnosis of Alzheimer's Disease (AD) and Mild Cognitive Impairment (MCI): Must meet the clinical diagnostic criteria for AD-related MCI and mild AD as defined by the National Institute on Aging and the Alzheimer's Association (NIA-AA) (2011); confirmed Aβ positivity through Aβ-PET/CT, Aβ-PET/MRI, or cerebrospinal fluid testing.
* MMSE ≥ 21 or MoCA ≥ 17 or CDR = 0.5
* No significant signs found in the neurological examination
* Participants must be capable of completing cognitive assessments and other tests.
* Informed consent must be obtained from the participants and their legal guardians, with a dated signature, prior to any operations or tests related to the protocol, committing to comply with the research procedures and cooperate throughout the study process.

Exclusion Criteria:

* Cognitive decline caused by other reasons: cerebrovascular disease, central nervous system infections, Creutzfeldt-Jakob disease, Huntington's disease, Parkinson's disease, Lewy body dementia, traumatic dementia, other physical and chemical factors (drugs, alcohol, CO, etc.), significant systemic diseases (hepatic encephalopathy, pulmonary encephalopathy, etc.), intracranial space-occupying lesions (subdural hematoma, brain tumor), endocrine system disorders (thyroid disease, parathyroid disease), and dementia caused by vitamin deficiencies or any other reasons.
* Patients with other unstable diseases, or those who have had a stroke or transient ischemic attack, bleeding disorders, or seizures within the previous 12 months.
* Patients with psychiatric disorders who meet DSM-IV criteria for schizophrenia or other mental illnesses, bipolar disorder, major depression, or delirium.
* Patients with unstable or severe heart, lung, liver, kidney, hematological diseases; those with known malignancies or other serious prognoses.
* Exclusion of cerebral amyloid angiopathy-related inflammation/β-amyloid-related cerebral vasculitis (CAAri/ABRA).
* Presence of uncorrectable visual or auditory impairments that prevent completion of relevant assessments or scales.
* Patients who cannot undergo MRI due to claustrophobia, pacemakers, defibrillators, or metal implants.
* MRI findings showing more than four microhemorrhages (diameter < 10 mm), evidence of surface iron deposition, vascular edema, diffuse white matter disease, multiple lacunar strokes, or any strokes involving major vascular regions. Presence of evidence of cerebral contusions, brain softening, cerebral aneurysms, or other vascular malformations, central nervous system (CNS) infections, as well as brain tumors other than meningiomas or arachnoid cysts.
* Patients taking warfarin, vitamin K antagonists, or direct oral anticoagulants (dabigatran, rivaroxaban, edoxaban, apixaban, betrixaban) or heparin; patients receiving thrombolysis; patients with coagulation disorders.
* Pregnant or lactating women.
* Patients deemed unsuitable for use by clinicians apart from the exclusion criteria listed above.
* Patients with severe allergies to lecanemab or any excipients of this product.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Renji Hospital, Shanghai Jiao Tong University School of Medicine Xuanwu Hospital, Capital Medical University Ruijin Hospital, Shanghai Jiao Tong University School of Medicine Shanghai Mental Health Center The First Affiliated Hospital, Zhejiang University School of Medicine The Second Affiliated Hospital of Guangzhou Medical University West China Hospital of Sichuan University Tianjin Medical University General Hospital Nantong First People's Hospital Huadong Hospital, Fudan University Jinhua Central Hospital Ningbo Second Hospital Nanjing Drum Tower Hospital Nanjing Brain Hospital The Affiliated Hospital of Guizhou Medical University
Sampling Method: Non-Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2025-03-13 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Chang of CDR-SB score | baseline, 9 month, 18 month
  CDR-SB, clinical dementia rating-sum of boxes

SECONDARY OUTCOMES:
Change of amyloid burden | baseline, 9 month, 18 month
  AV45-PET
Change of ADAS-cog score | baseline, 9 month, 18 month
  ADAS-cog, the Alzheimer's Disease Assessment Scale-Cognitive Subscale
Change of ADCS-ADL score | baseline, 9 month, 18 month
  ADCS-ADL, the Alzheimer's Disease Cooperative Study - Activities of Daily Living Scale (ADCS-ADL)
Change of MoCA score | baseline, 9 month, 18 month
  MoCA, the Montreal Cognitive Assessment
Change of BNT score | baseline, 9 month, 18 month
  BNT, the Boston Naming Test
Change of TMT score | baseline, 9 month, 18 month
  TMT, the trail making test
Change of HAMA and HAMD score | baseline, 9 month, 18 month
  HAMA, Hamilton Anxiety Scale; HAMD, Hamilton Depression Scale
Change of biomarkers | baseline, 9 month, 18 month
  p-tau181, p-tau217, Aβ40, Aβ42 , pEAβ3-42, GFAP, NFL, TRPC6 ( blood, urine, feces, gingival crevicular fluid, cerebrospinal fluid)
Positron emission tomography (PET) | baseline, 9 month, 18 month
  Other PET including FDG-PET, Tau-PET, TSPO-PET, SV2A-PET, exendin-4 (GLP-1R)-PET, colinergic receptor probe (ASEM) PET
Change of structural MRI | baseline, 9 month, 18 month
  3D T1-weighted, 3D T2-weighted and Diffusion Tensor Imaging (DTI)
Change of functional MRI | baseline, 9 month, 18 month
  Blood oxygenation level dependent (BOLD) imaging
Change of magnetic susceptibility | baseline, 9 month, 18 month
  Quantitative susceptibility mapping (QSM) imaging
Change of perfusion imaging | baseline, 9 month, 18 month
  Arterial spin labeling (ASL) imaging
Whole Genome Sequencing | baseline
Change of speech information | baseline, 9 month, 18 month
  Speech recording of Cookie-theft description task, using self-developed ASR speech analysis software (China software copyright number: 2016RS164680) for speech analysis

CONTACTS AND LOCATIONS:
Overall Officials: Gang Wang, Principal Investigator — RenJi Hospital
Locations (15):
- China (15):
  - Xuanwu Hospital, Capital Medical University, Beijing, China
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangdong, China
  - The Affiliated Hospital of Guizhou Medical University, Guizhou, China
  - Nanjing Brain Hospital, Jiangsu, China
  - Nanjing Drum Tower Hospital, Jiangsu, China
  - Nantong First People's Hospital, Jiangsu, China
  - Huadong Hospital, Fudan University, Shanghai, China
  - Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China
  - Shanghai Mental Health Center, Shanghai, China
  - West China Hospital of Sichuan University, Sichuan, China
  - Tianjin Medical University General Hospital, Tianjin, China
  - Jinhua Central Hospital, Zhejiang, China
  - Ningbo Second Hospital, Zhejiang, China
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No